CLINICAL TRIAL: NCT06494514
Title: A Single-center, Randomized, Interventional Controlled Study of NALIRIFOX Combined With PD-1 Sequential Radiotherapy Versus AG Combined With PD-1 Sequential Radiotherapy for First-line Treatment of Locally Advanced Pancreatic Cancer
Brief Title: NALIRIFOX Combined With PD-1 Sequential Radiotherapy Versus AG Combined With PD-1 Sequential Radiotherapy as First-line Treatment of Locally Advanced Pancreatic Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Du Juan (Other)
Responsible Party: Sponsor-Investigator, Du Juan, chief physician choice, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Organization: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-DEY-PC-JS02
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Locally Advanced Pancreatic Cancer
MeSH Terms: interventions — Gemcitabine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NALIRINOX combined with PD-1 synchronous sequential SBRT (Experimental): Nal-IRI+Oxaliplatin+5-FU +PD-1, these drugs are given on d1, d15, 28 days as one cycle, 6-8 cycles. SBRT is performed during the third cycle.
  Interventions: Drug: nal-IRI+Oxaliplatin+5-FU/LV+PD-1; Drug: Gemcitabine + albumin-paclitaxel+PD-1
- AG combined with PD-1 synchronous sequential SBRT (Experimental): Gemcitabine + albumin-paclitaxel +PD-1, these drugs are given on d1, d8, 21 days as one cycle, 6-8 cycles. SBRT is performed during the third cycle.
  Interventions: Drug: nal-IRI+Oxaliplatin+5-FU/LV+PD-1; Drug: Gemcitabine + albumin-paclitaxel+PD-1

INTERVENTIONS:
Drug: nal-IRI+Oxaliplatin+5-FU/LV+PD-1 — These drugs are given on d1, d15, 28 days as one cycle. 6-6 treatment cycles. SBRT is performed in third cycles.
Drug: Gemcitabine + albumin-paclitaxel+PD-1 — These drugs are given on d1, d8, 21 days as one cycle. 6-6 treatment cycles. SBRT is performed in third cycles.

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of NALIRINOX combined with PD-1 synchronous sequential SBRT or AG combined with PD-1 synchronous sequential SBRT as first line systematical therapy in patients with ocally advanced pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmed pancreatic cancer;
2. ECOG performance no more than 2;
3. Radiographically assessed as locally advanced pancreatic cancer according to NCCN guidelines;
4. No previous anti-tumor therapy；
5. Able and willing to provide a written informed consent;

Exclusion Criteria:

* 1. Prior anti-tumor therapy of any kind; 2. Severe infection (>NCI CTC grade 2); 3.Patients with autoimmune disease or immune deficiency who are treated with immunosuppressive drugs; 4.Patients with bleeding tendency; 5. Pregnant or lactating women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2027-04-01 (Estimated); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
mPFS | Up to 12 months
  Time from randomization to disease progression and/or death.

SECONDARY OUTCOMES:
mOS | Up to 24 months
  Time from randomization to death
ORR | Up to 12 months
  According to RECIST version 1.1, the proportion of patients who achieved remission (PR+CR) after treatment and maintained the minimum time-frame requirement.
DCR | Up to 12 months
  According to RECIST version 1.1, the proportion of patients who achieved remission (PR+CR) and stable lesion (SD) after treatment and maintained the minimum time-frame requirements.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School; Min Tu, Study Director — The First Affiliated Hospital with Nanjing Medical University
Locations (2):
- China (2):
  - FirstNanjingMU, Nanjing, Jiangsu
  - The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu